CLINICAL TRIAL: NCT00517465
Title: A Multi-center, Double-blind, Randomized, Placebo-controlled, Parallel-group, Multiple-ascending-dose Study to Investigate the Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of R1511 in Type 2 Diabetic (T2D) Patients
Brief Title: A Multiple Ascending Dose Study of R1511 in Patients With Type 2 Diabetes Mellitus.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NP20945
Record Dates: First submitted 2007-08-16; First posted 2007-08-17 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: RG1511
- 2 (Experimental)
  Interventions: Drug: RG1511
- 3 (Experimental)
  Interventions: Drug: RG1511
- 4 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — po bid
  Arms: 4
Drug: RG1511 — Starting multiple doses of 100mg po bid escalated in subsequent groups of patients to potential maximum multiple dose of 1200mg po bid.
  Arms: 1; 2; 3

SUMMARY:
This 4 arm study will evaluate the pharmacokinetics, pharmacodynamics, safety and tolerability of multiple ascending doses of R1511 compared to placebo in patients with type 2 diabetes mellitus. The starting dose of R1511 will be 100mg po bid for 5 1/2 days; this dose will be escalated in subsequent groups of patients to a potential maximum of 1200mg po bid for 5 1/2 days after a satisfactory assessment of blinded safety, tolerability, pharmacokinetic and pharmacodynamic data of the previous dose. The anticipated time on study treatment is <3 months, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-65 years of age;
* type 2 diabetic patients;
* naive to anti-diabetic therapy, or taken off current anti-diabetic therapy for >=2 weeks before first treatment.

Exclusion Criteria:

* type 1 diabetes mellitus;
* clinically significant cardiovascular disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2007-09; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
AEs, laboratory parameters, vital signs. | Throughout study
Glucose AUC | Days -1, 1 and 8.

SECONDARY OUTCOMES:
Insulin, C-peptide, glucagon and GLP-1 AUC | Days -1, 1 and 8
24h glucose | Days -1, 1 and 8
Lipid profiles | Days -1 and 8
Pharmacokinetic parameters | Days 1 and 8

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (7):
- Germany (2):
  - Berlin
  - Neuss
- Hungary (2):
  - Balatonfüred
  - Budapest
- Bratislava, Slovakia
- United Kingdom (2):
  - Slough
  - Welwyn Garden City